CLINICAL TRIAL: NCT02940717
Title: Clinical Evaluation of the Fracture Resistance for E-max Cad and Vita Suprinity Laminate Veneers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed mohamed osman Youssef, Internal resident at fixed prothodontics department faculty of oral and dental medicine cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: emax_vita
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Tooth Discoloration
MeSH Terms: conditions — Tooth Discoloration | interventions — VITA Suprinity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vita suprinity (Experimental): Vita Suprinity is a recent material with glass ceramic enriched with zirconia (approx. 10 % by weight) that offer practices and laboratories a high-strength, zirconia-reinforced lithium silicate ceramic (ZLS).
  Interventions: Other: Vita suprinity
- Emax cad (Active Comparator): lithium disilicate glass-ceramic which is etchable and proved to have good success rate if used for laminate venners
  Interventions: Other: Emax CAD

INTERVENTIONS:
Other: Vita suprinity — New glass ceramic material
  Other Names: zirconia-reinforced lithium silicate ceramic
  Arms: Vita suprinity
Other: Emax CAD — standard etchable glass ceramic used for laminate venneers
  Other Names: lithium disilicate glass ceramic
  Arms: Emax cad

SUMMARY:
Patients need laminate veneer for their teeth usually use Emax CAD as an etchable ceramic. Yet fracture may occur so a stronger material is needed. Vita Suprinity is a recent material with glass ceramic enriched with zirconia (approx. 10% by weight) that offer practices and laboratories a high-strength, zirconia-reinforced lithium silicate ceramic (ZLS) and can be used to fabricate laminate veneers but the investigators have to know clinically it is fracture resistance, so the investigators are going to have Parallel groups in a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

All subjects are required to be:

* From 18-60 years old, and able to read and sign the informed consent document.
* Physically and psychologically able to tolerate conventional restorative procedures
* Have no active periodontal or pulpal diseases, have teeth with good restorations
* Patients with teeth problems indicated for laminate veneer (e.g. discoloration, fracture not involve more than 50% enamel loss, mild malposition, ….)
* Willing to return for follow-up examinations and evaluation

Exclusion Criteria:

* Patients in the growth stage with partially erupted teeth
* Patient with fractured teeth of more than 50% enamel loss
* Patients with poor oral hygiene and motivation
* Pregnant women
* Psychiatric problems or unrealistic expectations
* Lack of opposite occluding dentition in the area intended for restoration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Fracture resistance assessed by clinical evaluation using dental mirror and probe according to the modified united states public health criteria | 1 Year
  clinical evaluation of Fracture resistance

SECONDARY OUTCOMES:
Patient satisfaction assessed using a Questionnaire | 1 Year
  Questionnaire for patient satisfaction

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elsaka SE, Elnaghy AM. Mechanical properties of zirconia reinforced lithium silicate glass-ceramic. Dent Mater. 2016 Jul;32(7):908-14. doi: 10.1016/j.dental.2016.03.013. Epub 2016 Apr 14. PMID 27087687
- [Background] Gresnigt MM, Kalk W, Ozcan M. Clinical longevity of ceramic laminate veneers bonded to teeth with and without existing composite restorations up to 40 months. Clin Oral Investig. 2013 Apr;17(3):823-32. doi: 10.1007/s00784-012-0790-5. Epub 2012 Jul 21. PMID 22821429
- [Background] Weyhrauch M, Igiel C, Scheller H, Weibrich G, Lehmann KM. Fracture Strength of Monolithic All-Ceramic Crowns on Titanium Implant Abutments. Int J Oral Maxillofac Implants. 2016 Mar-Apr;31(2):304-9. doi: 10.11607/jomi.4601. PMID 27004277